CLINICAL TRIAL: NCT05498558
Title: The Selection of Pregnancy for Patients After Tubal Ectopic Pregnancy Treatment In Pudong New Area
Brief Title: The Selection of Pregnancy for Patients After Tubal Ectopic Pregnancy Treatment
Acronym: TSOPFPATEPT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: Shanghai 7th People's Hospital (Other); Shanghai Zhoupu Hospital (Unknown); Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiFMIH2022-LSD
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Tubal-preserving Treatment of Tubal Ectopic Pregnancy; Tubal Pregnancy; Pregnancy Preparation
MeSH Terms: conditions — Pregnancy, Tubal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ovulation occurs on the healthy side: In tubal-presering patient who received treatment of tubal ectopic pregnancy,only when ovulation occurs on the healthy side of ovary,it may be considered to try to conceive; otherwise, contraception is recommended.
  Interventions: Other: No intervention.
- Ovulation occurs on the either side: In tubal-presering patient who received treatment of tubal ectopic pregnancy,ovulation occurs on the either side of ovary,it may be considered to try to conceive.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
The incidence of re-ectopic pregnancy in patients with tubal ectopic pregnancy increases significantly, which may be related to the condition of the fallopian tubes, such as tubal inflammation, tubal obstruction and other high-risk factors that may lead to tubal ectopic pregnancy; it is also associated with the treatment of the previous tubal ectopic pregnancy. Compared with salpingectomy, the treatment of preserving the fallopian tubes increased the incidence of re-ectopic pregnancy while increasing the pregnancy rate of the patient. For tubal-preserving patients, the most common option currently used is to recommend that monitoring ovulation during each menstrual cycle if they choose to conceive naturally rather than IVF. If ovulation occures on the healthy side of the ovary, it may be considered to try to conceive; Otherwise, contraception is recommended. However, there are uncertainties about this option. Based on this, we intend to conduct a multicenter clinical trial to verify the effectiveness of the ovulation preparation regimen on the healthy side of ovary.

DETAILED DESCRIPTION:
Tubal ectopic pregnancy is a disease that seriously affects women's physical and mental health and reproductive health, not only can there be some short-term complications such as rupture of tubal pregnancy and massive bleeding in the abdominal cavity, but also can lead to a decrease in female fertility, and the incidence of subsequent ectopic pregnancy has increased significantly. In recent years, with the development of diagnosis and treatment methods, the proportion of serious clinical events such as rupture of tubal pregnancy and massive hemorrhage in patients has decreased significantly. However, there is little research on the long-term damage of tubal pregnancy to women's fertility, especially how to avoid the occurrence of re-ectopic pregnancy, and there is no definitive and effective program.The incidence of re-ectopic pregnancy in patients with tubal ectopic pregnancy increases significantly, which may be related to the condition of the fallopian tubes, such as tubal inflammation, tubal obstruction and other high-risk factors that may lead to tubal ectopic pregnancy; it is also associated with the treatment of the previous tubal ectopic pregnancy. Compared with salpingectomy, the treatment of preserving the fallopian tubes increased the incidence of re-ectopic pregnancy while increasing the pregnancy rate of the patient.It is reported that the incidence of re-ectopic pregnancy in patients who choose salpingotomy is significantly higher than salpingectomy.Patients receiving conservative treatment and expectant treatment with methotrexate have a similar incidence of re-ectopic pregnancy as in patients receving salpingotomy.For tubal-preserving patients, the most common option currently used is to recommend that monitoring ovulation during each menstrual cycle if they choose to conceive naturally rather than IVF. If ovulation occures on the healthy side of the ovary, it may be considered to try to conceive; Otherwise, contraception is recommended. However, there are uncertainties about this option. Based on this, we intend to conduct a multicenter clinical trial to verify the effectiveness of the ovulation preparation program on the healthy side of ovary.We plan to randomly divide patients who meet the inclusion criteria into two groups:preparation for pregnancy in each ovulatory cycle and in healthy ovulatory cycle. Monitor the development of the patient's follicles each cycle, follow the patient to pregnancy, and analyze the patient's ovulation rate of healthy ovary, pregnancy rate, ectopic pregnancy rate and the time required from preparation to be pregnant, so as to determine whether the healthy side ovulation preparation program can improve the patient's normal pregnancy rate and reduce the ectopic pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

1. After tubal pregnancy treatment (including expectant therapy, medication, salpingotomy), the blood hCG value returns to normal;
2. The patient has fertility requirements;
3. The age of the patient is between 18-41 years old;
4. Regular menstruation;
5. There is no abnormality in the husband's semen examination;
6. No history of sex hormone drugs in the 3 months prior to the examination;
7. No underlying diseases such as heart, liver, kidneys and brain;
8. No history of tuberculosis;
9. Normal blood routine examination (WBC≥ 4*109/L, HB≥100g/L, PLT≥100*109/L);
10. Normal liver and kidney function tests;
11. Normal thyroid function;
12. The patient can withstand and receive follicle monitoring during pregnancy;
13. Negative for pregnancy test before treatment.

Exclusion Criteria:

1. Cervical pregnancy, cesarean scar pregnancy, cornual pregnancy, interstitial pregnancy;
2. The age of the patient < 18 years or > 41 years;
3. Irregular menstruation or abnormal results of sex hormone tests during follow-up;
4. Abnormal results of the man's semen examination during the follow-up period;
5. The patient has a tendency to bleed easily;
6. History of myometriosis and endometriosis;
7. Abnormal blood routine examination or liver and kidney function;
8. History of cardiovascular diseases, including severe hypertension, severe arrhythmias, history of myocardial infarction;
9. History of hepatitis B or C infection and patient has a detectable viral load;
10. Patients with active tuberculosis;
11. History of malignant tumors;
12. Unable to regularly monitor the follicles during pregnancy;
13. Unconditional long-term follow-up;

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with fertility needs who received tubal-preserving treatment during prior tubal ectopic pregnant in Shanghai First Maternity and Infant Hospital, Shanghai Zhoupu Hospital, Shanghai Seventh People's Hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of tubal pregnancy within12 months in both groups of patients. | 2023.10
  Tubal ectopic pregnancy refers to the implantation of embryo in the fallopian tubes.

SECONDARY OUTCOMES:
Rates of pregnancy and miscarriage within 12 months in both groups of patients. | 2023.10
  Clinical pregnancy is defined as ultrasound suggesting a gestational sac, with or without fetal heartbeat; miscarriage is defined as ultrasound suggesting that the fetus is inanimate or that the fetus has miscarried spontaneously.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan is undecided now.

REFERENCES:
- [Result] Mol F, van Mello NM, Strandell A, Strandell K, Jurkovic D, Ross J, Barnhart KT, Yalcinkaya TM, Verhoeve HR, Graziosi GCM, Koks CAM, Klinte I, Hogstrom L, Janssen ICAH, Kragt H, Hoek A, Trimbos-Kemper TCM, Broekmans FJM, Willemsen WNP, Ankum WM, Mol BW, van Wely M, van der Veen F, Hajenius PJ; European Surgery in Ectopic Pregnancy (ESEP) study group. Salpingotomy versus salpingectomy in women with tubal pregnancy (ESEP study): an open-label, multicentre, randomised controlled trial. Lancet. 2014 Apr 26;383(9927):1483-1489. doi: 10.1016/S0140-6736(14)60123-9. Epub 2014 Feb 3. PMID 24499812